CLINICAL TRIAL: NCT05630066
Title: A Phase IIa Multicenter, Open-label, 12-week Study to Investigate the Pharmacokinetics and Safety and to Provide Proof of Mechanism of Alogabat in Children and Adolescents Aged 5-17 Years With Angelman Syndrome (AS) With Deletion Genotype
Brief Title: A Study to Investigate the Pharmacokinetics (PK) and Safety and to Provide Proof of Mechanism of Alogabat in Children and Adolescents Aged 5-17 Years With Angelman Syndrome (AS) With Deletion Genotype.
Acronym: Aldebaran
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP41315; 2022-501844-14-00 (EU CTIS Number)
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Intervention Model Description: There will be up to 7 cohorts. The adolescents aged 15-17 will receive the adult dose. Dosing in Part 1 is pre-specified. Cohorts in Part 1 enroll a specific age range (15-17, 10-14, 5-9), with older cohorts being initiated prior to younger ones.
  Part 2 features mixed-age cohorts, with age-adjusted doses. Within each Part 2 cohort, two different doses of alogabat may be used: one up to Week 2 (Dose A), and the other from Week 3 to Week 12 (Dose B). Part 2 opens enrolment for ages 10-17 years following analysis of the 2-week data from the Part 1 cohorts aged 15-17 years and 10-14 years. Ages 5-9 years may enroll in Part 2 following analysis of the 2-week data from the Part 1 cohort with participants aged 5-9 years. Part 2 Cohort 2 will open enrollment across ages following the review of Week 2 and Week 4 data in Part 2 Cohort 1. A total of two optional cohorts may be utilized in this study, allocated to Part 1 and/or Part 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 Adult Alogabat Dose (Age 15-17) (Experimental): In Part 1 of the study participants will receive alogabat once a day (QD).
  Interventions: Drug: Alogabat
- Part 1 Age-adjusted Dose (Age 10-14) (Experimental): In Part 1 of the study, participants will receive age-adjusted QD doses of alogabat.
  Interventions: Drug: Alogabat
- Part 1 Age-adjusted Dose (Age 5-9) (Experimental): In Part 1 of the study, participants will receive age-adjusted QD doses of alogabat.
  Interventions: Drug: Alogabat
- Part 2 Cohort 1 (Experimental): In Part 2 of the study, the dosing will depend upon the results of Part 1 with two different dose levels per cohort. Doses can be age-adjusted.
  Interventions: Drug: Alogabat
- Part 2 Cohort 2 (Experimental): In Part 2 of the study, the dosing will depend upon the interim results with two different dose levels per cohort. Doses can be age-adjusted.
  Interventions: Drug: Alogabat
- Part 1 Optional Cohort (Experimental): If dose adjustments (e.g., increase or decrease in dose) are required, particularly due to uncertainty of the clearance estimates (e.g., due to high variability) or over-/underprediction of the pediatric clearance versus adult clearance, additional participants may be recruited in any of the of the 3 age-groups in order to confirm the exposure equivalence. A total of two optional cohorts may be utilized in this study, allocated to Part 1 and/or Part 2.
  Interventions: Drug: Alogabat
- Part 2 Optional Cohort (Experimental): In Part 2 of the study, the dosing will depend upon the interim results with two different dose levels per cohort. Doses can be age-adjusted.
  Interventions: Drug: Alogabat

INTERVENTIONS:
Drug: Alogabat — Alogabat will be administered QD with dose depending on cohort and age of the participant.

SUMMARY:
This is a two-part, Phase IIa, multicenter, 12-week, open-label study. Up to 56 participants with deletion AS aged 5-17 years (inclusive) will be enrolled in the study.

DETAILED DESCRIPTION:
The study will have Part 1-dose confirmations and Part 2 with dose levels to be decided based on the cumulative PK, electroencephalography (EEG), and safety data emerging from Part 1.

The dose levels for the first cohort of Part 2 will be decided based on the cumulative PK, EEG, and safety data emerging from Part 1.

Part 2 will explore the change in EEG beta-band power relative to baseline at Week 2, Week 4 (i.e., approximately 2 weeks after the start of the Dose B), and at the end of the 12-week treatment period after daily administration of alogabat.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AS and a genetic subtype of deletion on chromosome 15q11q13 confirmed by a historical molecular diagnosis
* The participant's general health status, in the context of the disease under study, allows them to participate in a clinical trial in the opinion of the investigator
* The reliability of sexual abstinence for male and/or female enrollment eligibility needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of preventing drug exposure
* Female participants:

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and non-childbearing or remain abstinent and/or Hormonal contraceptive methods must be supplemented

-Male participants: Male contraception is not required in this study because of the minimal seminal dose transmitted through sexual intercourse

Exclusion Criteria:

* A molecular diagnosis of AS with genotypic classification of any type besides the molecular diagnosis as specified in Inclusion Criterion
* Concurrent cardiovascular disease considered not well controlled by drug treatment, including participants with clinically significant hypertension, bradycardia and arrhythmias, myocardial infarction (MI) within 12 months of screening or uncompensated heart failure
* Confirmed clinically significant abnormality on 12-lead electrocardiogram (ECG), including:
* a QT corrected for heart rate using the Fridericia's correction factor (QTcF) of >/= 450 ms (based on the average of 3 consecutive measurements) for participants older than 10 years old
* a QT corrected for heart rate using Bazett's formula (QTcB) of >/= 450 ms (based on the average of 3 consecutive measurements) for participants up to, and including, the age of 10 years old
* Congenital heart diseases not treated and congenital QT corrected for heart rate (QTc) prolongation or family history of Long QT Syndrome
* Medical history of malignancy if not considered cured or if occurred within the last 5 years with the exception of fully excised non-melanoma skin cancers or in-situ carcinoma of the cervix that has been successfully treated
* Concomitant disease, condition, or treatment that would either interfere with the conduct of the study or pose an unacceptable risk to the participant in the opinion of the investigator
* Known active or uncontrolled bacterial, viral, or other infection (excluding fungal infections of nail beds) or any major episode of infection or hospitalization (relating to the completion of the course of antibiotics) within 6 weeks prior to the start of drug administration. Rescreening is allowed once the infection is cured and if the rescreening criteria are met
* Any concomitant condition that might interfere with the clinical evaluation of AS and that is not related to AS
* Known history of human immunodeficiency virus (HIV) or hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks of Screening or planned during the study. Rescreening is allowed not earlier than 12 weeks after the surgery and if the rescreening criteria are met.
* Use of prohibited medications within 6 weeks or 5 half-lives (t1/2) prior to start of study medication on Day 1 (whichever is longer)
* Clinically significant loss of blood within 3 months prior to screening defined by participant age and weight per recommendations from Duke University (2012)
* Any prior or current treatment with an investigational study drug within 6 weeks or 5 times the t1/2 of the investigational molecule (whichever is longer) prior to baseline or prior or current use of an investigational medical device within 6 weeks prior to baseline or if the device is still active. Concurrent or planned concurrent participation in any clinical study (including observational and non-interventional studies) without approval of the Investigator.
* Previous participation in a cellular therapy, gene therapy, or gene editing clinical study
* Clinically significant vital sign or ECG abnormalities at Screening
* Confirmed clinically significant abnormality in hematological, chemistry or coagulation laboratory parameters
* Uncorrected hypokalemia or hypomagnesaemia
* Positive test result at screening for hepatitis B surface antigen (HBsAg), HCV (untreated), or HIV-1/2. Participants with HCV who have been successfully treated and who test negative for HCV ribonucleic acid (HCV RNA) may be considered eligible for entry into the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Part 1: Age-group Based Ratio of Plasma PK Parameter, Area Under the Concentration-time Curve (AUC) | Up to 12 Weeks
  Age-group based ratio of plasma PK parameters in pediatric participants with AS versus data collected from adult healthy volunteers and participants with autism spectrum disorder (ASD) (AUC)
Part 1: Age-group Based Ratio of Plasma PK Parameter, Apparent Clearance (CL/F) | Up to 12 Weeks
  Age-group based ratio of plasma PK parameters in pediatric participants with AS versus data collected from adult healthy volunteers and participants with ASD (CL/F)
Part 2: Change From Baseline to Week 2, 4, and 12 in Resting State EEG Power in the Beta Band | Week 2, 4, and 12

SECONDARY OUTCOMES:
Parts 1 and 2: Plasma PK Parameter of Alogabat, Maximum Concentration (Cmax) | Up to 12 Weeks
  Plasma PK parameter of alogabat Cmax as derived using a population-pharmacokinetic (popPK) model
Parts 1 and 2: Plasma PK Parameter of Alogabat, AUC | Up to 12 Weeks
  Plasma PK parameter of alogabat AUC as derived using a popPK model
Parts 1 and 2: Plasma PK Parameter of Alogabat, CL/F | Up to 12 Weeks
  Plasma PK parameter of alogabat CL/F derived using a popPK model
Parts 1 and 2: Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 18 Weeks
  Incidence and severity of AEs and SAEs
Parts 1 and 2: Incidence of Treatment Discontinuations due to AEs | Up to 18 Weeks
  Incidence of treatment discontinuations due to AEs
Parts 1 and 2: Incidence of Daytime Sleepiness Assessed With the Karolinska Sleepiness Scale (KSS), and Incidence of Sudden Onset of Sleep Assessed With Somnolence Diary | Up to 12 Weeks
  Incidence of daytime sleepiness assessed with the KSS, and incidence of sudden onset of sleep assessed with somnolence diary.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (6):
  - Rush Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Carolina Institute for Development DisabilitiesUniversity of North Carolina/School of Medicine, Carrboro, North Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Multicare Institute for Research and Innovation, Tacoma, Washington
- Queensland Children?s Hospital, South Brisbane, Queensland, Australia
- France (4):
  - CHRU de Brest, Brest
  - CHU Dijon Bourgogne Hôpital François Mitterand, Dijon
  - Hopital la Timone Enfants, Marseille
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Dr. Von Haunersches Kinderspital, München, Germany
- Italy (3):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - IRCCS Istituto G. Gaslini, Genoa, Liguria
  - IRCCS Eugenio Medea, Conegliano Veneto (TV), Veneto
- Spain (4):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat · Barcelona, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario de Navarra;Unidad de Neuropediatría, Pamploa, Navarre
  - Hospital Universitario Puerta De Hierro Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing
Supporting Information: Study Protocol